CLINICAL TRIAL: NCT03850405
Title: Effects of Dark Chocolate on Gut Microbiome and Cholesterol Reduction in Subjects With Moderate Dyslipidemia
Brief Title: Dark Chocolate, Cholesterol and Microbiota
Acronym: CHOCO-diet
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, piero portincasa, Professor of Medicine, Head Division of Internal Medicine, University of Bari
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1419UO
Record Dates: First submitted 2019-02-11; First posted 2019-02-21 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Dyslipidemias; Hypertriglyceridemia
MeSH Terms: conditions — Dyslipidemias; Hypertriglyceridemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chocolate (Experimental): 20 patients (matched per gender) undergoing a diet which includes 25g of dark chocolate (70%), i.e. ca. 145 kcal per day
  Interventions: Dietary Supplement: Dark Chocolate
- Control (No Intervention): 20 patients (matched per gender) undergoing a low-fat dietary regimen

INTERVENTIONS:
Dietary Supplement: Dark Chocolate — 20 patients (10 male, 10 female) will undergo a diet containing 25g of dark chocolate (70%), corresponding to ca. 145 kcal which will be detracted from the total caloric intake.
  Arms: Chocolate

SUMMARY:
Scientific evidence shows that a major consume of flavonoids is associated with a minor risk of coronary disease and a modification of the gut microbiome profile.

Dark chocolate has a major quantity of flavonoids by weight in comparison to wine, dark tea, blueberry juice, apples and, in particular the flavanols (i.e. catechin, epicatechin and procyanidin) can have protective and metabolic effects with reduction of the insulin resistance and improvement of the endothelial function in adults.

In line with the aforementioned evidence, the present study has the aim of analyze the effect of dark chocolate (70%) on cardiovascular risk and on the metabolism in a population with mild dyslipidemia.

DETAILED DESCRIPTION:
Chocolate, the main product deriving from cocoa beans (Theobroma cacao, from the Greek "food of the gods") has its origin in Mexico, where Maya, Inca and Aztecs practiced their cultivation. For centuries, it has been appreciated for its pleasant taste and for its beneficial effects on health, and it is one of the most sought-after worldwide, with a consumption greatly increasing in recent years thanks to a wide availability of products on the market.

Dietary choices are strongly influenced by the taste and consistency of foods. Fat is largely responsible for the sensory properties of many foods and, therefore, contribute greatly to the pleasure of eating. Dark chocolate consists of ≈43% of lipids, mainly represented by cocoa butter, the latter consisting on average of 33% of oleic acid, 25% of palmitic acid and 33% of stearic acid. Another component of chocolate is polyphenols, in particular flavonoids, substances with numerous beneficial effects for health, including antihypertensive, anti-inflammatory, antithrombotic, metabolic and prebiotic activity, playing a role in the change of human intestinal microbiota.

Recent scientific studies show an inverse correlation between flavonoid intake in the diet and the incidence of diabetes, such as to hypothesize the use of flavonoid-rich foods as potential nutritional supplements in the management of diabetes. The cocoa flavonoids can bring benefits to the insulin-resistance condition by improving endothelial function, modifying glucose metabolism and reducing oxidative stress, which is considered the main cause of insulin resistance. In healthy individuals and patients with moderate cardiovascular risk, regular flavonoid intake improves levels of cardiovascular biomarkers, lowering serum LDL cholesterol and triglycerides and increasing HDL cholesterol. The flavonoids present in cocoa can also inhibit platelet aggregation by down-regulation of the cellular synthesis of eicosanoids.

ELIGIBILITY:
Inclusion Criteria:

* Individuals able to fill an Informed Consent
* Aged 40-60 years old with 1:1 matched criteria, age difference of ± 1 year old
* Patients with mild dyslipidemia (total cholesterol 201-250 mg/dL, LDL≥155 mg/dL) with or without hypertriglyceridemia (150-180 mg/dL) who accept to be inserted in a program aimed to reduce their caloric intake, including diet alone or diet plus chocolate

Exclusion Criteria:

* Missing Informed Consent
* Diagnosis of organic diseases, including neoplastic inflammatory diseases or cardiovascular diseases
* Patients on statin therapy
* Drugs which can affect the gastrointestinal tract and interfere with the symptoms
* Pregnancy
* Presence of diseases with a prognosis of less than 12 months
* Hypersensitivity to chocolate or chocolate components

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2019-07-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Total Cholesterol | Baseline
  Total cholesterol in mg/100ml will be measured by serum extraction from 3ml of whole peripheral blood.
Triglycerides | Baseline
  Triglycerides in mg/dl will be measured by serum extraction from 3ml of whole peripheral blood.
HDL Cholesterol | Baseline
  HDL Cholesterol in mg/dl will be measured by serum extraction from 3ml of whole peripheral blood.
Counts of viable fecal bacterial cells | Baseline
  Estimate of microbial Shannon's (H') diversity from 3g faecal sample:
  Heterotrophic aerobic and anaerobic bacteria Total anaerobes Lactic acid bacteria Lactobacillus Lactococcus and Streptococcus Staphylococcus Bacteroides Porphyromonas and Prevotella Enterobacteria Aeromonas and Pseudomonas Bifidobacterium Enterococci

CONTACTS AND LOCATIONS:
Overall Officials: Piero Portincasa, MD, PhD, Principal Investigator — Clinica Medica "A. Murri", DIMO - University of Bari
Locations (1):
- Department of Biomedical Sciences Human Oncology - Clinica Medica "A. Murri", Bari, BA, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Latif R. Chocolate/cocoa and human health: a review. Neth J Med. 2013 Mar;71(2):63-8. PMID 23462053
- [Background] Shah SR, Alweis R, Najim NI, Dharani AM, Jangda MA, Shahid M, Kazi AN, Shah SA. Use of dark chocolate for diabetic patients: a review of the literature and current evidence. J Community Hosp Intern Med Perspect. 2017 Sep 19;7(4):218-221. doi: 10.1080/20009666.2017.1361293. eCollection 2017 Oct. PMID 29181133
- [Background] Schroeter H, Heiss C, Balzer J, Kleinbongard P, Keen CL, Hollenberg NK, Sies H, Kwik-Uribe C, Schmitz HH, Kelm M. (-)-Epicatechin mediates beneficial effects of flavanol-rich cocoa on vascular function in humans. Proc Natl Acad Sci U S A. 2006 Jan 24;103(4):1024-9. doi: 10.1073/pnas.0510168103. Epub 2006 Jan 17. PMID 16418281
- [Background] Ueshima K. Magnesium and ischemic heart disease: a review of epidemiological, experimental, and clinical evidences. Magnes Res. 2005 Dec;18(4):275-84. PMID 16548143
- [Background] Allen RR, Carson L, Kwik-Uribe C, Evans EM, Erdman JW Jr. Daily consumption of a dark chocolate containing flavanols and added sterol esters affects cardiovascular risk factors in a normotensive population with elevated cholesterol. J Nutr. 2008 Apr;138(4):725-31. doi: 10.1093/jn/138.4.725. PMID 18356327
- [Background] Hayek N. Chocolate, gut microbiota, and human health. Front Pharmacol. 2013 Feb 7;4:11. doi: 10.3389/fphar.2013.00011. eCollection 2013. No abstract available. PMID 23405053
- [Background] Davinelli S, Corbi G, Righetti S, Sears B, Olarte HH, Grassi D, Scapagnini G. Cardioprotection by Cocoa Polyphenols and omega-3 Fatty Acids: A Disease-Prevention Perspective on Aging-Associated Cardiovascular Risk. J Med Food. 2018 Oct;21(10):1060-1069. doi: 10.1089/jmf.2018.0002. Epub 2018 May 3. PMID 29723102
- [Background] Lee Y, Berryman CE, West SG, Chen CO, Blumberg JB, Lapsley KG, Preston AG, Fleming JA, Kris-Etherton PM. Effects of Dark Chocolate and Almonds on Cardiovascular Risk Factors in Overweight and Obese Individuals: A Randomized Controlled-Feeding Trial. J Am Heart Assoc. 2017 Nov 29;6(12):e005162. doi: 10.1161/JAHA.116.005162. PMID 29187388